CLINICAL TRIAL: NCT03665415
Title: Engaging Children With Mental Health and Developmental Disabilities and Their Parents to Adopt a Healthy Lifestyle: Piloting the Game Squad Home Exergaming & Virtual Health Coaching Intervention
Brief Title: Expanded Game Squad for Neurodiverse Youth
Acronym: NDGameSquad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merrimack College (Other)
Collaborators: University of Massachusetts, Worcester (Other); Pennington Biomedical Research Center (Other); Boston Medical Center Developmental and Behavioral Pediatrics Clinic (Unknown); Marblehead Public Schools (Unknown)
Responsible Party: Principal Investigator, April Bowling, Assistant Professor, Merrimack College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-FY18-19-1
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Physical Activity; Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Health Behavior; Developmental Disorder
MeSH Terms: conditions — Motor Activity; Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Health Behavior; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The project will be carried out in three phases: 1) Formative research to implement the intervention with n=6 youth in order to make any modifications necessary before embarking on the full pilot in both sites in the next phase; 2) The pilot intervention comprised of a randomized wait-list controlled pilot intervention at two sites (school and clinic) during the school year; 3) an unsupported follow up period where participants in the school-based intervention will be offered the intervention during the summer months without school staff support. Wait-listed school site participants will also receive the unsupported intervention in this phase.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded to assignment. Objective outcomes (physical activity, height, weight, blood pressure) will be collected by masked assessors. The primary investigator and all data analysts will be blinded to participant assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formative (Other): This stage represents an initial formative phase to implement the NDGame Squad intervention with small samples of youth in order to make any modifications necessary before embarking on the full pilot in both sites in the next phase. Three (n=3) participants from the school site only will participate in an initial 4-week Game Squad intervention in the first formative phase. Participant feedback including barriers to engagement and suggestions for improvements will be obtained via parent/caregiver and child interviews post-intervention.
  Interventions: Behavioral: NDGameSquad
- Pilot Intervention (Experimental): Participants in the pilot intervention arm will receive either 10 or 14 weeks of the NDGameSquad intervention. School site participants will receive 10 weeks during the school year, followed by another 4 weeks during summer vacation. Clinic site participants will receive 10 weeks only.
  Interventions: Behavioral: NDGameSquad
- Pilot Waitlist Control (Other): Participants at both sites randomized to the waitlist control arm will be asked to maintain current physical activity levels during the first 10-week period. They will then be provided the intervention equipment and training. School site control arm participants will then participate in a 4-week, unsupported summer NDGame Squad intervention. Clinic site control arm participants will not be required to participate in the NDGameSquad intervention.
  Interventions: Behavioral: NDGameSquad

INTERVENTIONS:
Behavioral: NDGameSquad — The intervention will be delivered within participants' homes. Participants will be provided a gaming console and exergames. Participants will be encouraged to meet a goal of 60 minutes/day of MVPA for the duration of the intervention by playing the exergames at least three times per week and engaging in non-screen based physical activity on other days. Participants will receive a booklet that includes a curriculum for playing weekly challenges. Participants will wear a FitBit during their exergaming sessions. Participants and parents meet bi-weekly with a health coach via video-chat using the exergame console. Sessions will identify and encourage specific physical activity, healthy eating, and healthy sleep habits. At the school site, participants will receive additional check-ins, engagement support, and health curricula from classroom teachers during the first 10 weeks of the intervention.

SUMMARY:
The proposed study will pilot the use of an adapted Game Squad intervention aimed at improving physical activity and other important health behaviors (nutrition, sleep hygiene, screen time habits) for children and adolescents receiving special education supports for behavioral health challenges, or who are served by the Boston Medical Center Developmental and Behavioral Pediatrics (BMC-DBP) clinic.

DETAILED DESCRIPTION:
The significant health disparities that exist among people with mental health conditions (MH) and developmental disabilities (DD), including autism spectrum disorder (ASD), have been documented through research and clinical practice. The majority of studies have focused on adults with these conditions, but due to the efforts of agencies such as the Maternal Child Health Bureau, the health disparities experienced by youth with MH and DD are increasingly recognized. These youth are more likely to be overweight and obese than their typically developing (TD) counterparts, have higher cardio-metabolic risk factors, and have lower levels of health-related fitness. These conditions can be partly attributed to the low physical activity levels and poor diet quality that have been observed in these populations. Multiple barriers that operate at the individual, community, and societal levels limit opportunities for these youth to achieve good health, and thus there is an urgent need for health promotion interventions to address these disparities. One novel way to address these barriers is to explore the use of virtual methods adapted specifically for this population to reach these children and families in their homes, while also investigating viable venues through which such interventions can be delivered and supported if necessary.

This study seeks to pilot a virtual health coaching and exercise program aimed at addressing modifiable lifestyle factors that can lead to improved health and well-being for youth with MH and DD. The Game Squad Home Exergaming program, originally developed by the Pennington Biomedical Research Center, is a theoretically-guided and evidence-based intervention that has shown effectiveness at engaging parents and children with overweight/obesity in regular physical activity and virtual health counseling. Game Squad utilizes home exergaming consoles (i.e., Kinect for Xbox video games that require physical activity for gameplay) for both caregiver and child exercise sessions, as well as to deliver virtual health counseling sessions to participants. These virtual health counseling sessions were aimed at improving non-exergame related physical activity. Importantly, during a recent RCT involving a socio-economically and racially diverse population over a six-month period, the intervention yielded clinically significant reductions in BMI z-score and cardiovascular disease risk factors, as well as increased moderate to vigorous physical activity (MVPA).

The proposed project seeks to determine whether the Game Squad intervention is acceptable and engaging to children and adolescents with MH and DD, adapt the health counseling sessions to encompass additional health behaviors and meet the needs of this population, as well as to assess feasibility of implementation through both a school-based program and a specialized clinic for children with MH/DD. This is achieved through innovative partnerships with several key collaborators: Merrimack College; the Pennington Biomedical Research Center; the Therapeutic Intervention Designed for Educational Success Program (TIDES) program, a public school special education collaborative in several north shore communities in Massachusetts; and the developmental-behavioral pediatrics clinic at Boston Medical Center (BMC-DBP), a clinical site associated with the MCHB-funded Developmental Pediatrics Research Network (DBP-NET).

ELIGIBILITY:
Inclusion Criteria:

* Receiving services either through the BMC-DBP or TIDES programs
* Wi-Fi and TV available in their home environment

Exclusion Criteria:

* Intellectual disability
* Chronic or physically disabling conditions for which strenuous physical activity is contra-indicated or not feasible

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline 7-day Actigraph MVPA after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Change in moderate to vigorous physical activity measured via hip-worn Actigraph accelerometer

SECONDARY OUTCOMES:
Change from baseline BMI after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Child body mass index change
Change from baseline blood pressure after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Child systolic and diastolic blood pressure change
Change from baseline parent perceptions of child health habits after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Change in parent report of child sleep, meal-time, screen and physical activity behaviors
Change from baseline child anxiety symptoms after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Change in parent and child reported Screen for Childhood Anxiety Related Emotional Disorder (SCARED) questionnaire. The full scale range is 0-82, with five sub-scales (panic disorder range 0-26; generalized anxiety disorder range 0-18; separation anxiety disorder range 0-16; social anxiety disorder range 0-14; school avoidance range 0-8). Higher score values indicate greater experience of symptoms. Total score is the sum of all sub-scores.
Change in child depression symptoms after 10 weeks of intervention | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Change in child reported modified Patient Health Questionnaire for Adolescents (PHQ-A) questionnaire, which assesses symptoms of depression. The scale has a total score range of 0-27 and there are no sub-scales. Greater values indicate greater experience of symptoms.
Change in child video game use habits | Collected within 14 days of intervention start (baseline) and end (follow-up after 10 week intervention)
  Change in child reported video game use questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Medical Center Developmental and Behavioral Pediatrics Clinic, Boston, Massachusetts
  - Marblehead Public Schools, Marblehead, Massachusetts

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Background] Anderson SE, Must A, Curtin C, Bandini LG. Meals in Our Household: reliability and initial validation of a questionnaire to assess child mealtime behaviors and family mealtime environments. J Acad Nutr Diet. 2012 Feb;112(2):276-84. doi: 10.1016/j.jada.2011.08.035. PMID 22741169
- [Background] Baglioni C, Nanovska S, Regen W, Spiegelhalder K, Feige B, Nissen C, Reynolds CF, Riemann D. Sleep and mental disorders: A meta-analysis of polysomnographic research. Psychol Bull. 2016 Sep;142(9):969-990. doi: 10.1037/bul0000053. Epub 2016 Jul 14. PMID 27416139
- [Background] Barnett A, Cerin E, Baranowski T. Active video games for youth: a systematic review. J Phys Act Health. 2011 Jul;8(5):724-37. doi: 10.1123/jpah.8.5.724. PMID 21734319
- [Background] Biddiss E, Irwin J. Active video games to promote physical activity in children and youth: a systematic review. Arch Pediatr Adolesc Med. 2010 Jul;164(7):664-72. doi: 10.1001/archpediatrics.2010.104. PMID 20603468
- [Background] Blaine B. Does depression cause obesity?: A meta-analysis of longitudinal studies of depression and weight control. J Health Psychol. 2008 Nov;13(8):1190-7. doi: 10.1177/1359105308095977. PMID 18987092
- [Background] Bowling A, Slavet J, Miller DP, Haneuse S, Beardslee W, Davison K. Cybercycling Effects on Classroom Behavior in Children With Behavioral Health Disorders: An RCT. Pediatrics. 2017 Feb;139(2):e20161985. doi: 10.1542/peds.2016-1985. Epub 2017 Jan 9. PMID 28069663
- [Background] Broder-Fingert S, Brazauskas K, Lindgren K, Iannuzzi D, Van Cleave J. Prevalence of overweight and obesity in a large clinical sample of children with autism. Acad Pediatr. 2014 Jul-Aug;14(4):408-14. doi: 10.1016/j.acap.2014.04.004. PMID 24976353
- [Background] Brown SA. Measuring perceived benefits and perceived barriers for physical activity. Am J Health Behav. 2005 Mar-Apr;29(2):107-16. doi: 10.5993/ajhb.29.2.2. PMID 15698978
- [Background] Cook BG, Li D, Heinrich KM. Obesity, Physical Activity, and Sedentary Behavior of Youth With Learning Disabilities and ADHD. J Learn Disabil. 2015 Nov-Dec;48(6):563-76. doi: 10.1177/0022219413518582. Epub 2014 Jan 21. PMID 24449262
- [Background] Cortese S, Morcillo Penalver C. Comorbidity between ADHD and obesity: exploring shared mechanisms and clinical implications. Postgrad Med. 2010 Sep;122(5):88-96. doi: 10.3810/pgm.2010.09.2205. PMID 20861592
- [Background] TRUE Consortium. Recommended standards for assessing blood pressure in human research where blood pressure or hypertension is a major focus. J Hum Hypertens. 2017 Aug;31(8):487-490. doi: 10.1038/jhh.2017.10. Epub 2017 Apr 13. No abstract available. PMID 28406234
- [Background] Davis C, Levitan RD, Smith M, Tweed S, Curtis C. Associations among overeating, overweight, and attention deficit/hyperactivity disorder: a structural equation modelling approach. Eat Behav. 2006 Aug;7(3):266-74. doi: 10.1016/j.eatbeh.2005.09.006. Epub 2005 Oct 17. PMID 16843230
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] Gao Z, Chen S, Pasco D, Pope Z. A meta-analysis of active video games on health outcomes among children and adolescents. Obes Rev. 2015 Sep;16(9):783-94. doi: 10.1111/obr.12287. Epub 2015 May 6. PMID 25943852
- [Background] Gariepy G, Nitka D, Schmitz N. The association between obesity and anxiety disorders in the population: a systematic review and meta-analysis. Int J Obes (Lond). 2010 Mar;34(3):407-19. doi: 10.1038/ijo.2009.252. Epub 2009 Dec 8. PMID 19997072
- [Background] Howard AL, Robinson M, Smith GJ, Ambrosini GL, Piek JP, Oddy WH. ADHD is associated with a "Western" dietary pattern in adolescents. J Atten Disord. 2011 Jul;15(5):403-11. doi: 10.1177/1087054710365990. Epub 2010 Jul 14. PMID 20631199
- [Background] Lee EC, Whitehead AL, Jacques RM, Julious SA. The statistical interpretation of pilot trials: should significance thresholds be reconsidered? BMC Med Res Methodol. 2014 Mar 20;14:41. doi: 10.1186/1471-2288-14-41. PMID 24650044
- [Background] Li SH, Jin XM, Shen XM, Wu SH, Jiang F, Yan CH, Yu XD, Qiu YL. [Development and psychometric properties of the Chinese version of Children's Sleep Habits Questionnaire]. Zhonghua Er Ke Za Zhi. 2007 Mar;45(3):176-80. Chinese. PMID 17504618
- [Background] Manu P, Dima L, Shulman M, Vancampfort D, De Hert M, Correll CU. Weight gain and obesity in schizophrenia: epidemiology, pathobiology, and management. Acta Psychiatr Scand. 2015 Aug;132(2):97-108. doi: 10.1111/acps.12445. Epub 2015 May 27. PMID 26016380
- [Background] Mazurek MO, Sohl K. Sleep and Behavioral Problems in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Jun;46(6):1906-1915. doi: 10.1007/s10803-016-2723-7. PMID 26823076
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Newcomer JW, Hennekens CH. Severe mental illness and risk of cardiovascular disease. JAMA. 2007 Oct 17;298(15):1794-6. doi: 10.1001/jama.298.15.1794. No abstract available. PMID 17940236
- [Background] O'Neil A, Quirk SE, Housden S, Brennan SL, Williams LJ, Pasco JA, Berk M, Jacka FN. Relationship between diet and mental health in children and adolescents: a systematic review. Am J Public Health. 2014 Oct;104(10):e31-42. doi: 10.2105/AJPH.2014.302110. PMID 25208008
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Peng W, Lin JH, Crouse J. Is playing exergames really exercising? A meta-analysis of energy expenditure in active video games. Cyberpsychol Behav Soc Netw. 2011 Nov;14(11):681-8. doi: 10.1089/cyber.2010.0578. Epub 2011 Jun 13. PMID 21668370
- [Background] Puyau MR, Adolph AL, Vohra FA, Zakeri I, Butte NF. Prediction of activity energy expenditure using accelerometers in children. Med Sci Sports Exerc. 2004 Sep;36(9):1625-31. PMID 15354047
- [Background] Rimmer JH, Rowland JL, Yamaki K. Obesity and secondary conditions in adolescents with disabilities: addressing the needs of an underserved population. J Adolesc Health. 2007 Sep;41(3):224-9. doi: 10.1016/j.jadohealth.2007.05.005. PMID 17707291
- [Background] Sechrist KR, Walker SN, Pender NJ. Development and psychometric evaluation of the exercise benefits/barriers scale. Res Nurs Health. 1987 Dec;10(6):357-65. doi: 10.1002/nur.4770100603. PMID 3423307
- [Background] Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: prevalence, comorbidity, and associated factors in a population-derived sample. J Am Acad Child Adolesc Psychiatry. 2008 Aug;47(8):921-9. doi: 10.1097/CHI.0b013e318179964f. PMID 18645422
- [Background] Staiano AE, Beyl RA, Guan W, Hendrick CA, Hsia DS, Newton RL Jr. Home-based exergaming among children with overweight and obesity: a randomized clinical trial. Pediatr Obes. 2018 Nov;13(11):724-733. doi: 10.1111/ijpo.12438. Epub 2018 Jul 20. PMID 30027607
- [Background] Strimas R, Davis C, Patte K, Curtis C, Reid C, McCool C. Symptoms of attention-deficit/hyperactivity disorder, overeating, and body mass index in men. Eat Behav. 2008 Dec;9(4):516-8. doi: 10.1016/j.eatbeh.2008.07.005. Epub 2008 Aug 8. PMID 18928919
- [Background] Trost SG, Pate RR, Freedson PS, Sallis JF, Taylor WC. Using objective physical activity measures with youth: how many days of monitoring are needed? Med Sci Sports Exerc. 2000 Feb;32(2):426-31. doi: 10.1097/00005768-200002000-00025. PMID 10694127
- [Derived] Bowling AB, Slavet J, Hendrick C, Beyl R, Nauta P, Augustyn M, Mbamalu M, Curtin C, Bandini L, Must A, Staiano AE. The Adaptive GameSquad Xbox-Based Physical Activity and Health Coaching Intervention for Youth With Neurodevelopmental and Psychiatric Diagnoses: Pilot Feasibility Study. JMIR Form Res. 2021 May 14;5(5):e24566. doi: 10.2196/24566. PMID 33988508